CLINICAL TRIAL: NCT01458990
Title: Proton Pump Inhibitors and Dysbiosis in Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jasmohan Bajaj, Associate Professor, Hunter Holmes Mcguire Veteran Affairs Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BAJAJ004
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Cirrhosis; Healthy
MeSH Terms: conditions — Fibrosis | interventions — Omeprazole

STUDY DESIGN:
Intervention Model Description: PPI withdrawal (decompensated patients only) and PPI initiation (compensated and decompensated patients)
Oversight: Data Monitoring Committee: No

ARMS (2):
- PPI inititation (Experimental): Adding 40mg omeprazole QD for 14 days
  Interventions: Drug: Omeprazole
- PPI withdrawal (Active Comparator): The intervention here is systematically withdrawing chronic PPI for 14 days
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Omeprazole — 20mg PO BID for 20 days

SUMMARY:
The purpose of this study is to find out whether the use of medications that suppress acid in your stomach can change the composition of your bowel bacteria.

ELIGIBILITY:
Inclusion Criteria for PPI initiation study:

* Cirrhosis not on current PPI or acid suppressive therapy
* No systemic antibiotics or probiotics

Exclusion Criteria for PPI initiation study:

* On systemic antibiotics
* On PPI or acid suppression therapy already
* unable to give informed consent
* Allergy to proton pump inhibitors

Inclusion Criteria for PPI withdrawal study:

* Cirrhosis on current PPI for an FDA-unapproved indication
* No systemic antibiotics or probiotics

Exclusion Criteria for PPI withdrawal study:

* On systemic absorbable antibiotics
* On PPI or acid suppression therapy for an FDA-approved indication
* unable to give informed consent
* unwilling to withdraw PPI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-10; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bajaj JS, Cox IJ, Betrapally NS, Heuman DM, Schubert ML, Ratneswaran M, Hylemon PB, White MB, Daita K, Noble NA, Sikaroodi M, Williams R, Crossey MM, Taylor-Robinson SD, Gillevet PM. Systems biology analysis of omeprazole therapy in cirrhosis demonstrates significant shifts in gut microbiota composition and function. Am J Physiol Gastrointest Liver Physiol. 2014 Nov 15;307(10):G951-7. doi: 10.1152/ajpgi.00268.2014. Epub 2014 Sep 25. PMID 25258407
- [Derived] Pena Rodriguez M, Fagan A, Sikaroodi M, Gillevet PM, Bajaj JS. Proton Pump Inhibitor Use and Complications of Cirrhosis Are Linked With Distinct Gut Microbial Bacteriophage and Eukaryotic Viral-Like Particle Signatures in Cirrhosis. Clin Transl Gastroenterol. 2024 Feb 1;15(2):e00659. doi: 10.14309/ctg.0000000000000659. PMID 37937851
- [Derived] Bajaj JS, Thacker LR, Fagan A, White MB, Gavis EA, Hylemon PB, Brown R, Acharya C, Heuman DM, Fuchs M, Dalmet S, Sikaroodi M, Gillevet PM. Gut microbial RNA and DNA analysis predicts hospitalizations in cirrhosis. JCI Insight. 2018 Mar 8;3(5):e98019. doi: 10.1172/jci.insight.98019. PMID 29515036
- [Derived] Bajaj JS, Liu EJ, Kheradman R, Fagan A, Heuman DM, White M, Gavis EA, Hylemon P, Sikaroodi M, Gillevet PM. Fungal dysbiosis in cirrhosis. Gut. 2018 Jun;67(6):1146-1154. doi: 10.1136/gutjnl-2016-313170. Epub 2017 Jun 3. PMID 28578302

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from McGuire VAMC hepatology clinics
Period: Overall Study
Arm/Group | PPI Inititation | PPI Withdrawal
Started | 45 | 15
Completed | 45 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PPI Inititation | PPI Withdrawal | Total
Number analyzed (Participants) | 45 | 15 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 14 | 54
  >=65 years | 5 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (7.6) | 59 (6.7) | 58 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 42 | 14 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 6 | 22
  White | 29 | 9 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 45 | 15 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Overgrowth of Oral Microbiota in Their Stool After PPI Therapy Withdrawal or Initiation
Description: Analysis at baseline will be compared to that at 2 weeks using Multitagged sequencing. Number of patients with overgrowth of oral microbiota in their stool after PPI therapy withdrawal or initiation were specifically analyzed.
Time Frame: 2 weeks
Population: Comparison were made between groups on/off PPI therapy using Linear discriminant analysis effect size (LEFSe) and using the Quantitative Insights Into Microbial Ecology (QIIME) pipeline and also the relative proportion (%) of oral-origin microbiota were studied
Measure: Count of Participants; unit: Participants
Arm/Group | PPI Inititation | PPI Withdrawal
Number analyzed (Participants) | 45 | 15
Participants | 45 | 15

2. Secondary Outcome: Number of Patients With Adverse Events During Initiation or Withdrawal of PPI Therapy
Description: Analysis at baseline will be compared to that at 2 weeks. This will be specifically, changes in those with PPI withdrawal compared to those with PPI initiation
Time Frame: 2 weeks
Population: No safety or tolerability issues were seen during the study
Measure: Count of Participants; unit: Participants
Groups:
- PPI Initiation; PPI Withdrawal: No safety signals were identified
Arm/Group | PPI Initiation | PPI Withdrawal
Number analyzed (Participants) | 45 | 15
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: During study period of 14 days
Description: Standard definitions used
Arm/Group | PPI Inititation | PPI Withdrawal
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/15
Other Adverse Events (participants affected / at risk) | 0/45 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT01458990/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT01458990/SAP_001.pdf